CLINICAL TRIAL: NCT03647891
Title: The Impact of Early Diagnosis and Treatment of Obstructive Sleep Apnea on Hospital Readmission in Hospitalized Cardiac Patients: the CV Readmit Clinical Trial
Brief Title: Impact of Early Diagnosis and Treatment of OSA on Hospital Readmission in Hospitalized Cardiac Patients
Acronym: CV Readmit
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study on hold
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Dennis Hwang, MD, Medical Director, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPSleep-003
Record Dates: First submitted 2017-01-06; First posted 2018-08-27 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: OSA; Heart Failure; Myocardial Infarction; Arrhythmia, Cardiac
Keywords: obstructive sleep apnea; CPAP; hospital readmission; heart failure; myocardial infarction; cardiac arrhythmia
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Arrhythmias, Cardiac; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CPAP Intervention Pathway (Experimental): Patients will receive continuous positive airway pressure (CPAP) therapy in the hospital followed by home CPAP therapy. Their home CPAP therapy will include wireless connectivity, which includes adherence data. Furthermore, the patients will be entered into our usual automated platform (USleep; ResMed Corp) in which patients with suboptimal CPAP use will be sent messages (based on patient preference) in order to ensure adherence to therapy. This platform is already a standard part of our usual care.
  The patients will receive CPAP in addition to contemporary standard of care pharmacotherapy for their underlying cardiac condition(s). They will follow up at the Fontana Sleep Center within 1 month after discharge for assessment of CPAP use and asked to complete a questionnaire packet. Patients will be followed during the 30-day period and assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms.
  Interventions: Device: Continuous Positive Airway Pressure
- Usual Care Pathway (No Intervention): Patients will receive contemporary standard of care pharmacotherapy for their underlying cardiac condition(s) and will not receive CPAP therapy for the duration of the study. They will be asked to follow up at the Fontana Sleep Center within 1 month after discharge for a repeat outpatient portable sleep study and asked to complete a questionnaire packet. The results of the outpatient portable sleep studies will be compared with the in-patient portable sleep study. Patients will also be asked to follow up with the Fontana Sleep Center within 1 month after discharge for assessment of primary and secondary outcomes. Patients will be followed during the 30-day period and assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — CPAP is an FDA approved therapy machine for patients diagnosed with OSA. CPAP provides positive air pressure to the patients throat to ensure the patients airway stays open during sleep. CPAP is the gold standard treatment for OSA, but there is limited research that demonstrates whether or not CPAP can improve clinical outcomes in patients with cardiovascular disease. Therefore, our investigators plan to initiate CPAP therapy in patients hospitalized for cardiovascular disease to investigate whether there is an improvement in cardiac function and clinical outcomes (e.g. mortality).
  Other Names: CPAP; APAP
  Arms: CPAP Intervention Pathway

SUMMARY:
The purpose of this study is to determine whether early diagnosis of obstructive sleep apnea and initiation of and adherence to CPAP therapy in hospitalized cardiac patients would impact 30-day hospital readmission rates.

DETAILED DESCRIPTION:
Study investigators have designed a single-center, randomized control trial to evaluate the impact of early diagnosis and treatment of obstructive sleep apnea (OSA) in hospitalized cardiac patients on hospital readmission, symptoms, and healthcare utilization. This study targets a high risk population (hospitalized cardiac patients) and targets early initiation of continuous positive airway pressure (CPAP) therapy in patients diagnosed with OSA. Investigators intend to enroll all consenting participants hospitalized with a primary cardiac diagnosis, which include congestive heart failure, arrhythmia's, and acute coronary syndromes. The study is unique and the answer to its question - whether early diagnosis of OSA and initiation of and adherence to CPAP therapy in hospitalized cardiac patients will reduce 30-day readmission rates - is unknown. The objective is twofold: to improve quality of care and decrease preventable hospitalizations through early diagnosis and implementation of this early diagnosis and intervention model for this subset of patients may slow progression of cardiac disease, offset a large public health and financial burden, and improve overall outcomes.

Study investigators believe that the study, which involves human subjects, is in accordance with general ethical principles. It should be noted that diagnosis and subsequent treatment of OSA during hospitalization is not part of routine practice, and that the control group truly would follow "usual care". Moreover, patients who are deemed very sick (as outlined in the exclusion criteria) will be excluded from the study. Finally, half of enrolled participants will receive early CPAP therapy which may potentially benefit those patients beyond what is currently "usual care".

Study Design

The study is a single-center, randomized control trial designed to evaluate the impact of early diagnosis and treatment of obstructive sleep apnea (OSA) in hospitalized cardiac patients on hospital readmission, symptoms, and healthcare utilization. Consecutive patients who meet inclusion criteria hospitalized with a primary diagnosis of heart failure, arrhythmia, or acute coronary syndrome will be asked to participate in the study. Patients who agree and sign consent will undergo a portable sleep study to diagnose OSA-predominant sleep disordered breathing. Patients will also complete a questionnaire packet consisting of the following standardized questionnaires: sleep history questionnaire, Epworth Sleepiness Scale (ESS), EQ5D-5L, and PROMIS questionnaire. Each patient who meets inclusion criteria and consents to the study will undergo an inpatient portable sleep study (ApneaLink, Resmed Corp). This is a Type III study which is an unattended study that measures nasal pressure, respiratory effort, oxygen saturation, and body position. A study investigator will apply the portable device, and a board-certified sleep medicine physician (co-investigators) will interpret these studies. The study will be performed while the patient is on room air (not on oxygen), thus the study may not be applied on the first hospitalized night (if oxygen therapy is required), but delayed until the patient is appropriate to be off oxygen.

A diagnosis of OSA will be made if the apnea-hypopnea index with 4% oxygen desaturation is greater than 5 (AHI4%≥5) with at least 50% of events consistent with obstructive rather than central physiology. Study participants with OSA will then be randomized into one of two pathways: Intervention Pathway and Usual Care Pathway.

Intervention Pathway Patients will receive CPAP therapy in the hospital followed by home CPAP therapy. A sleep center respiratory therapy/sleep technologist case manager will perform a bedside mask fit, CPAP education, and set up their outpatient follow-up appointments with the sleep center. Their home CPAP therapy will be a loaner from the sleep medicine department that includes wireless connectivity so that adherence data is available to the investigators throughout the duration of the study. Furthermore, the patients will be entered into our usual automated platform (USleep; ResMed Corp) in which patients with suboptimal CPAP use will be sent messages (email or text based on patient preference) in order to ensure adherence to therapy. This platform is already a standard part of our usual care.

The patients will receive CPAP in addition to the contemporary standard of care pharmacotherapy for their underlying cardiac condition(s). They will be asked to follow up at the Fontana Sleep Center within 1 month after discharge for assessment of CPAP use and asked to complete the aforementioned questionnaire packet (with the exception of the STOP BANG questionnaire). During the appointment, the sleep center will troubleshoot CPAP use when appropriate; otherwise, requests for additional troubleshooting will be at the discretion of the patient (as is currently our usual care). In addition, patients will receive a $50 stipend for participation in the study. Patients will be assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms at the 1-month period

Usual Care Pathway Patients will receive contemporary standard of care pharmacotherapy for their underlying cardiac condition(s) and will not receive CPAP therapy for the duration of the study. They will be asked to follow up at the Fontana Sleep Center within 1 month after discharge for a repeat outpatient portable sleep study and asked to complete the aforementioned questionnaire packet (with the exception of the STOP BANG questionnaire). The results of the outpatient portable sleep studies will be compared with the in-patient portable sleep study. At the one-month follow up appointment, patients will receive a $50 stipend for participation in the study. Patients will be assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms at the 1-month period

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente member
* Males or female, any race, and age 18 and older
* OSA-predominant (AHI at or above 5) sleep disordered breathing
* Primary diagnosis upon admission of congestive heart failure, acute coronary syndrome, or arrhythmias
* Congestive heart failure (Acute or acute on chronic systolic heart failure, Acute or acute on chronic diastolic heart failure)
* Acute coronary syndrome (ST segment elevation myocardial infarction, Non-ST segment myocardial infarction, Unstable angina)
* Arrhythmias (Tachyarrhythmias, Atrial fibrillation, Atrial flutter, Bradyarrhythmias, Sinus bradycardia, 2nd degree atrioventricular block, Complete heart block)
* Appropriate to perform portable sleep study while on room air (no oxygen)
* Patients who are able and willing to give informed consent

Exclusion Criteria:

* Use of CPAP within 6 months of enrollment
* Patients with CSA-predominant sleep disordered breathing
* Patients who are "sleepy": ESS at or above 11
* Commercial driver's license or other occupational hazards (operating heavy machinery)
* Non-English speaking (validated questionnaires are currently limited to English)
* Patients with chronic respiratory failure requiring oxygen therapy or non-invasive ventilation.
* Patients requiring tracheostomy
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Hospital readmission | 30 days
  Number of occasions patient has been admitted to the hospital
Mortality rates | 30 days
  Number of patients who have died

SECONDARY OUTCOMES:
Clinic and urgent care visits | 30 days
  Appointments with any medical providers (sleep, cardiac, primary) at a clinic or urgent care facility
Off work orders | 30 days
  Note from provider ordering/requesting patient to be dismissed from work for medical reasons (sick, injured, etc.)
STOP BANG | 30 days
  Snoring, tiredness, observed apnea, blood pressure, body mass index, age, neck circumference, and gender (STOP BANG) is the name of a OSA screening questionnaire. Questionnaire contains 8 "Yes/No" questions and the number of "Yes" answers provide a total score (range 0-8). Scores of at least 3 are typically considered to indicate risk of OSA.
Epworth Sleepiness Scale (ESS) | 30 days
  Epworth Sleepiness Scale measures degree of sleepiness. 8 scenarios are described and the responder indicates their likelihood of dozing unintentionally (range 0-3). A total of the scores are added (range 0-24) and typically scores of at least 11 indicate excessive sleepiness.
EQ5D-5L | 30 days
  EuroQoL 5-dimension 5-level measures health-related quality of life that can be used for wide range of health conditions. The questionnaire consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The patients can rate each dimension based on 5 level severity scale: no problems, slight problems, moderate problems, severe problems and extreme problems.This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
PROMIS | 30 days
  Patient Reported Outcome Measurement Information System is a 10 item questionnaire that measures physical, mental, and social health in adults. It can be used on the general population and patients with chronic conditions. Patients rate their health based on a severity scale of 1-5 (1 indicates poor health) and the scoring system allows each question/item to be evaluated separately.
Comparing inpatient portable monitor versus 30-day follow up portable monitor results in usual care group | 30 days
  Evaluating the change of sleep diagnostic test results from the hospital to 1-month after being discharged (only for patients enrolled in the Usual Care pathway)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hwang, MD, Principal Investigator — Fontana Medical Center, Kaiser Permanente
Locations (1):
- Sleep Center; San Bernardino County Medical Center, Kaiser Permanente, Fontana, California, United States